CLINICAL TRIAL: NCT01858363
Title: Prospective, Randomized, Multi-center, Single-blinded Study for the Treatment of Subjects Presenting With De Novo Occluded/Stenotic or Re-occluded/Restenotic Lesions of the Superficial Femoral or Popliteal Arteries Using Paclitaxel or Bare Percutaneous Transluminal Angioplasty Balloon Catheter
Brief Title: ILLUMENATE EU Randomized Clinical Trial
Acronym: EU RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TP 1360
Record Dates: First submitted 2013-05-08; First posted 2013-05-21 (Estimated); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Arterial Disease; Claudication
Keywords: Peripheral arterial disease; claudication; drug-coated balloon; drug-eluting balloon
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel-coated balloon (Experimental): Subjects with de novo occluded/stenotic or re-occluded/restenotic lesions will be randomly assigned to treatment with a Paclitaxel-coated balloon or bare balloon.
  Interventions: Device: CVI Paclitaxel-coated Percutaneous Transluminal Angioplasty Balloon Catheter
- Bare balloon (Placebo Comparator): Subjects with de novo occluded/stenotic or re-occluded/restenotic lesions will be randomly assigned to treatment with a Paclitaxel-coated balloon or bare balloon.
  Interventions: Device: Bare Percutaneous Transluminal Angioplasty Balloon Catheter

INTERVENTIONS:
Device: CVI Paclitaxel-coated Percutaneous Transluminal Angioplasty Balloon Catheter
  Arms: Paclitaxel-coated balloon
Device: Bare Percutaneous Transluminal Angioplasty Balloon Catheter
  Arms: Bare balloon

SUMMARY:
This is a prospective, randomized, multi-center, single-blind study to demonstrate the safety and effectiveness of the CVI Paclitaxel-coated percutaneous transluminal angioplasty (PTA) balloon versus bare PTA balloon for the treatment of patients with de novo occluded/stenotic or reoccluded/restenotic lesions of the superficial femoral (SFA) and popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic leg ischemia requiring treatment of the superficial femoral or popliteal arteries
* Rutherford clinical category 2, 3 or 4
* Male or non-pregnant female at least 18 years

Exclusion Criteria:

* Co-existing clinically significant aneurismal disease of the abdominal aorta, iliac or popliteal arteries
* Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy
* Known intolerance of study medications, paclitaxel or contrast agent
* Active participation in another investigational device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schroeder, M.D., Principal Investigator — Center for Diagnostic Radiology & Minimally Invasive Therapy, The Jewish Hospital
Locations (1):
- Center for Diagnostic Radiology and Minimally Invasive Therapy, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schroeder H, Werner M, Meyer DR, Reimer P, Kruger K, Jaff MR, Brodmann M; ILLUMENATE EU RCT Investigators. Low-Dose Paclitaxel-Coated Versus Uncoated Percutaneous Transluminal Balloon Angioplasty for Femoropopliteal Peripheral Artery Disease: One-Year Results of the ILLUMENATE European Randomized Clinical Trial (Randomized Trial of a Novel Paclitaxel-Coated Percutaneous Angioplasty Balloon). Circulation. 2017 Jun 6;135(23):2227-2236. doi: 10.1161/CIRCULATIONAHA.116.026493. Epub 2017 Apr 19. PMID 28424223
- [Result] Brodmann M, Werner M, Meyer DR, Reimer P, Kruger K, Granada JF, Jaff MR, Schroeder H; ILLUMENATE EU RCT Investigators. Sustainable Antirestenosis Effect With a Low-Dose Drug-Coated Balloon: The ILLUMENATE European Randomized Clinical Trial 2-Year Results. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2357-2364. doi: 10.1016/j.jcin.2018.08.034. PMID 30522663
- [Derived] Lyden SP, Brodmann M, Parikh SA, Krishnan P, Schroeder H, Werner M, Holden A, Ouriel K, Tarra T, Gray WA. Four-year patient-level pooled mortality analysis of the ILLUMENATE US Pivotal and EU randomized controlled trials. J Vasc Surg. 2022 Feb;75(2):600-607. doi: 10.1016/j.jvs.2021.07.244. Epub 2021 Sep 8. PMID 34506898
- [Derived] Gray WA, Jaff MR, Parikh SA, Ansel GM, Brodmann M, Krishnan P, Razavi MK, Vermassen F, Zeller T, White R, Ouriel K, Adelman MA, Lyden SP. Mortality Assessment of Paclitaxel-Coated Balloons: Patient-Level Meta-Analysis of the ILLUMENATE Clinical Program at 3 Years. Circulation. 2019 Oct;140(14):1145-1155. doi: 10.1161/CIRCULATIONAHA.119.040518. Epub 2019 Sep 30. PMID 31567024

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Lesions
Groups:
- Paclitaxel-coated Balloon: Subjects with de novo occluded/stenotic or re-occluded/restenotic lesions will be randomly assigned to treatment with a Paclitaxel-coated balloon or bare balloon.
  CVI Paclitaxel-coated Percutaneous Transluminal Angioplasty Balloon Catheter
- Bare Balloon: Subjects with de novo occluded/stenotic or re-occluded/restenotic lesions will be randomly assigned to treatment with a Paclitaxel-coated balloon or bare balloon.
  Bare Percutaneous Transluminal Angioplasty Balloon Catheter
Period: Overall Study
Arm/Group | Paclitaxel-coated Balloon | Bare Balloon
Started | 222; 254 Lesions | 72; 79 Lesions
Pre-discharge Visit | 219; 251 Lesions | 72; 79 Lesions
1-month Visit | 214; 246 Lesions | 68; 75 Lesions
6-month Visit | 208; 239 Lesions | 64; 71 Lesions
12-month Vist | 205; 235 Lesions | 61; 67 Lesions
24-month Visit | 184; 209 Lesions | 58; 64 Lesions
36-month Visit | 169; 194 Lesions | 53; 59 Lesions
48-month Visit | 157; 179 Lesions | 53; 59 Lesions
Completed | 146; 167 Lesions | 46; 51 Lesions
Not Completed | 76; 87 Lesions | 26; 28 Lesions
Not completed — Death | 35 | 9
Not completed — Withdrawal by Subject | 28 | 14
Not completed — Lost to Follow-up | 13 | 3

BASELINE CHARACTERISTICS:
Population: The Baseline Participants are based on the Intent-to-Treat (ITT) analysis set. The safety data for the adverse events section will be based on the Safety Set which has 219 participants in the Paclitaxel-coated arm and 68 in the Bare balloon arm.
Units Other Than Participants: lesions
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel-coated Balloon | Bare Balloon | Total
Number analyzed (Participants) | 222 | 72 | 294
Number analyzed (lesions) | 254 | 79 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.2) | 69.0 (8.6) | 67.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 23 | 85
  Male | 160 | 49 | 209
Rutherford Clinical Category [Count of Participants; unit: Participants] — The Rutherford-Becker Clinical Categories (RCC) are a classification system of chronic limb ischemia ranging from 0 (asymptomatic; no hemodynamically significant occlusive disease) to 6 (major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable). Lower categories represent better clinical status. Population: The Rutherford Clinical Category assessment was missing for 1 Paclitaxel-coated Balloon patient and for 1 Bare Balloon patient.
  Participants
    number analyzed (Participants) | 221 | 71 | 292
    Rutherford Clinical Category 2 | 34 | 15 | 49
    Rutherford Clinical Category 3 | 183 | 55 | 238
    Rutherford Clinical Category 4 | 4 | 1 | 5
Diabetes [Count of Participants; unit: Participants] | 83 | 26 | 109
Hypertension [Count of Participants; unit: Participants] | 173 | 60 | 233
Hyperlipidemia [Count of Participants; unit: Participants] | 137 | 49 | 186
Smoking status [Count of Participants; unit: Participants]
  Never Smoked | 24 | 12 | 36
  Previous or current | 198 | 60 | 258
Baseline Ankle Brachial Index [Mean (Standard Deviation); unit: ratio] — The Ankle-Brachial Index (ABI) is calculated ratio of the highest ankle blood pressure to the highest arm blood pressure. The ABI is a non-invasive tool for screening for Peripheral Artery Disease. Population: The ABI is part of the most missed assessments at baseline which accounts for the missing data. For some participants, ABI is non-measurable or the number too high suggesting non-compressible vessels (with a pressure cuff) and thus cannot be reported.
  ratio
    number analyzed (Participants) | 212 | 68 | 280
    (all) | 0.72 (0.21) | 0.69 (0.26) | 0.71 (0.22)
Lesion length (mm) [Mean (Standard Deviation); unit: mm] — Population: For 3 Paclitaxel-coated Balloon subjects, the Core Laboratory considered the treated area as 1 lesion instead of 2 lesions as reported by the sites.
  For 1 lesion, the Core Laboratory could only assess lesion location and calcification based on available images (All other baseline lesion characteristics are missing).
  mm
    number analyzed (lesions) | 250 | 79 | 329
    (all) | 71.8 (51.9) | 70.8 (52.7) | 71.6 (52.0)
Lesion type [Count of Units; unit: lesions]
  De novo | 234 | 71 | 305
  Restonotic | 20 | 8 | 28
Total Occlusion [Count of Units; unit: lesions] — Population: For 3 Paclitaxel-coated Balloon subjects, the Core Laboratory considered the treated area as 1 lesion instead of 2 lesions as reported by the sites.
  For 1 lesion, the Core Laboratory could only assess lesion location and calcification based on available images (All other baseline lesion characteristics are missing).
  lesions
    number analyzed (lesions) | 250 | 79 | 329
    (all) | 48 | 15 | 63
Calcification [Count of Units; unit: lesions] — Population: For 3 Paclitaxel-coated Balloon subjects, the Core Laboratory considered the treated area as 1 lesion instead of 2 lesions as reported by the sites.
  For 1 lesion, the Core Laboratory could only assess lesion location and calcification based on available images (All other baseline lesion characteristics are missing).
  lesions
    number analyzed (lesions) | 251 | 79 | 330
    None/Mild | 140 | 47 | 187
    Moderate | 79 | 24 | 103
    Severe | 32 | 8 | 40
Diameter stenosis [Mean (Standard Deviation); unit: % Diameter Stenosis] — Diameter stenosis is calculated as the difference between the minimal luminal diameter (MLD) from the target reference vessel diameter (RVD), divided by the RVD, and multiplied by 100 to get the percentage of stenosis. The RVD is typically calculated by averaging the MLD of the healthy part of the vessel both proximal and distal to the vessel lesion Population: For 3 Paclitaxel-coated Balloon subjects, the Core Laboratory considered the treated area as 1 lesion instead of 2 lesions as reported by the sites.
  For 1 lesion, the Core Laboratory could only assess lesion location and calcification based on available images (All other baseline lesion characteristics are missing).
  % Diameter Stenosis
    number analyzed (lesions) | 250 | 79 | 329
    (all) | 78.7 (16.0) | 80.8 (15.7) | 79.2 (15.9)
Reference vessel Diameter [Mean (Standard Deviation); unit: mm] — Population: For 3 DCB subjects, the Core Laboratory considered the treated area as 1 lesion instead of 2 lesions as reported by the sites.
  For 1 lesion, the Core Laboratory could only assess lesion location and calcification based on avalaible images (All other baseline lesion characterics are missing).
  mm
    number analyzed (lesions) | 250 | 79 | 329
    (all) | 5.02 (0.79) | 4.77 (0.69) | 4.96 (0.78)
# of patent run-off vessels [Count of Participants; unit: Participants] — Population: The lesions characterics are reported as analyzed by angiographic core laboratory by quantitative angiography.
  Participants
    number analyzed (Participants) | 211 | 68 | 279
    0 | 18 | 4 | 22
    1 | 40 | 9 | 49
    2 | 68 | 31 | 99
    3 | 85 | 24 | 109
pre-dilatation performed [Count of Units; unit: lesions] | 254 | 78 | 332
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women. Population: BMI data was not available for 4 participants in the Paclitaxel-coated balloon group.
  kg/m^2
    number analyzed (Participants) | 218 | 72 | 290
    (all) | 27.2 (4.7) | 27.8 (4.7) | 27.3 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Patency at 12-months
Description: The primary efficacy endpoint was patency at 12 months post-procedure defined as the absence of target lesion restenosis determined by duplex ultrasound peak systolic velocity ratio (PSVR) ≤2.5 and freedom from clinically-driven target lesion revascularization (CD-TLR).
Time Frame: 12 months
Population: The analysis for the primary patency was based on the lesion success and not participant success. In the Paclitaxel-coated balloon arm, 222 subjects represents 254 lesions. Of those 254 lesions, only 224 lesions were evaluable. In the Bare balloon arm, 72 subjects represents 79 lesions. Of those 79 lesions, only 66 lesions were evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Paclitaxel-coated Balloon | Bare Balloon
Number analyzed (Participants) | 222 | 72
Number analyzed (lesions) | 224 | 66
percentage of lesions | 83.9 [78.5 to 88.5] | 60.6 [47.8 to 72.4]

2. Primary Outcome: Percentage of Patients With Freedom From Device and Procedure Related Target Limb Major Amputation or Death Through 30-days Post-procedure and Clinically-driven Target Lesion Revascularization at 12-month
Description: The primary safety endpoint was freedom from device and procedure-related death through 30 days post-procedure and freedom from target limb major amputation and clinically-driven target lesion revascularization (CD-TLR) through 12 months post-procedure.
Time Frame: 30-Days and 12-Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel-coated Balloon | Bare Balloon
Number analyzed (Participants) | 222 | 72
percentage of participants | 94.1 [90.0 to 96.9] | 83.3 [71.5 to 91.7]

ADVERSE EVENTS:
Time Frame: The adverse events presented were collected through 12 Months. The data presented is based off the Safety Set (analysis set). The Safety Set excludes 7 participants who were not treated with a study device.
Arm/Group | Paclitaxel-coated Balloon | Bare Balloon
All-Cause Mortality (participants affected / at risk) | 35/219 | 9/68
Serious Adverse Events (participants affected / at risk) | 118/219 | 38/68
Other Adverse Events (participants affected / at risk) | 180/219 | 51/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel-coated Balloon (N=219) | Bare Balloon (N=68)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 2 (2) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (3) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 2 (2) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 9 (11) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
ENDOCARDIAL FIBROELASTOSIS (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 1 (1) | 1 (1)
EYELID PTOSIS (Eye disorders) | 1 (1) | 0 (0)
LENS DISLOCATION (Eye disorders) | 0 (0) | 1 (1)
MACULAR DEGENERATION (Eye disorders) | 2 (2) | 0 (0)
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 (0) | 2 (5)
PROCTITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
CATHETER SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0)
CATHETER SITE HAEMORRHAGE (General disorders) | 5 (5) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
DEVICE OCCLUSION (General disorders) | 4 (4) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3 (3) | 0 (0)
IMPAIRED HEALING (General disorders) | 0 (0) | 1 (1)
NECROSIS (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0)
THROMBOSIS IN DEVICE (General disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 0 (0) | 1 (2)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (3) | 0 (0)
PNEUMONIA (Infections and infestations) | 3 (3) | 0 (0)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
TUBERCULOSIS OF GENITOURINARY SYSTEM (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CONFUSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL REOCCLUSION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 6 (6) | 12 (13)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
TENDON INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
BLOOD GLUCOSE FLUCTUATION (Investigations) | 1 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FACET JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
POLYCYTHAEMIA VERA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
ATAXIA (Nervous system disorders) | 0 (0) | 1 (1)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 6 (7) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2) | 0 (0)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
MIGRAINE WITH AURA (Nervous system disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
BLADDER MASS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CAROTID ENDARTERECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
CARPAL TUNNEL DECOMPRESSION (Surgical and medical procedures) | 1 (1) | 0 (0)
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 2 (2) | 0 (0)
GASTROINTESTINAL DILATION PROCEDURE (Surgical and medical procedures) | 1 (1) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
PERIPHERAL ENDARTERECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
BLUE TOE SYNDROME (Vascular disorders) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
FEMORAL ARTERY DISSECTION (Vascular disorders) | 17 (18) | 6 (6)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 5 (6) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 4 (4) | 0 (0)
INTERMITTENT CLAUDICATION (Vascular disorders) | 3 (3) | 1 (1)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 3 (3) | 0 (0)
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 3 (3) | 1 (1)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 15 (20) | 6 (9)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0)
PERIPHERAL EMBOLISM (Vascular disorders) | 2 (2) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel-coated Balloon (N=219) | Bare Balloon (N=68)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
EOSINOPHILIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 3 (3) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 4 (4) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (3) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 3 (4) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 10 (14) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
ENDOCARDIAL FIBROELASTOSIS (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
CERUMEN IMPACTION (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 1 (1) | 1 (2)
CHORIORETINOPATHY (Eye disorders) | 1 (1) | 0 (0)
DIABETIC RETINOPATHY (Eye disorders) | 1 (1) | 0 (0)
EYELID PTOSIS (Eye disorders) | 1 (1) | 0 (0)
LENS DISLOCATION (Eye disorders) | 0 (0) | 1 (1)
MACULAR DEGENERATION (Eye disorders) | 2 (2) | 0 (0)
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (1)
VITREOUS HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 5 (6) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (2) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 (0) | 2 (5)
PROCTITIS (Gastrointestinal disorders) | 1 (2) | 0 (0)
SALIVARY GLAND CYST (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTH DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
CATHETER SITE HAEMATOMA (General disorders) | 4 (4) | 2 (2)
CATHETER SITE HAEMORRHAGE (General disorders) | 7 (7) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
DEVICE BREAKAGE (General disorders) | 1 (1) | 0 (0)
DEVICE OCCLUSION (General disorders) | 4 (5) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3 (3) | 0 (0)
IMPAIRED HEALING (General disorders) | 1 (1) | 1 (1)
LOCAL SWELLING (General disorders) | 1 (1) | 0 (0)
LOCALISED OEDEMA (General disorders) | 1 (1) | 0 (0)
NECROSIS (General disorders) | 1 (2) | 1 (1)
OEDEMA (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 5 (5) | 1 (1)
PAIN (General disorders) | 1 (1) | 0 (0)
PUNCTURE SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0)
THROMBOSIS IN DEVICE (General disorders) | 1 (1) | 0 (0)
BILIARY CIRRHOSIS PRIMARY (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLESTASIS (Hepatobiliary disorders) | 0 (0) | 1 (2)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
LIVER DISORDER (Hepatobiliary disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 8 (8) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0)
PERITONITIS (Infections and infestations) | 1 (3) | 0 (0)
PNEUMONIA (Infections and infestations) | 3 (3) | 1 (1)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 1 (1)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
TUBERCULOSIS OF GENITOURINARY SYSTEM (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONFUSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
NECK INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PERIPHERAL ARTERIAL REOCCLUSION (Injury, poisoning and procedural complications) | 4 (4) | 3 (4)
PERIPHERAL ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 20 (20) | 15 (21)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
SEROMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TENDON INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANKLE BRACHIAL INDEX DECREASED (Investigations) | 3 (3) | 0 (0)
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD COUNT ABNORMAL (Investigations) | 1 (1) | 0 (0)
BLOOD GLUCOSE FLUCTUATION (Investigations) | 1 (2) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 1 (1)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 14 (14) | 5 (7)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (10) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FACET JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (3)
OSTEOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 14 (15) | 4 (4)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SINUS TARSI SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADRENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
POLYCYTHAEMIA VERA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
ATAXIA (Nervous system disorders) | 0 (0) | 1 (1)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 8 (10) | 1 (1)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 2 (2)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2) | 0 (0)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 3 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
MIGRAINE WITH AURA (Nervous system disorders) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
SENSORY LOSS (Nervous system disorders) | 1 (1) | 0 (0)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1)
BLADDER MASS (Renal and urinary disorders) | 1 (1) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 0 (0)
URGE INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 3 (3) | 0 (0)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BLISTER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CAROTID ENDARTERECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
CARPAL TUNNEL DECOMPRESSION (Surgical and medical procedures) | 1 (1) | 0 (0)
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 2 (2) | 0 (0)
GASTROINTESTINAL DILATION PROCEDURE (Surgical and medical procedures) | 1 (1) | 0 (0)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
MOLE EXCISION (Surgical and medical procedures) | 1 (1) | 0 (0)
PERIPHERAL ENDARTERECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0)
ANGIODYSPLASIA (Vascular disorders) | 1 (1) | 0 (0)
BLUE TOE SYNDROME (Vascular disorders) | 1 (2) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
FEMORAL ARTERY DISSECTION (Vascular disorders) | 21 (22) | 7 (7)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 7 (9) | 1 (1)
HAEMATOMA (Vascular disorders) | 4 (4) | 1 (1)
HYPERTENSION (Vascular disorders) | 3 (3) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 4 (4) | 0 (0)
INTERMITTENT CLAUDICATION (Vascular disorders) | 15 (15) | 3 (4)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 0 (0)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 4 (5) | 0 (0)
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 3 (3) | 1 (1)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 21 (29) | 9 (21)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 2 (3) | 0 (0)
PERIPHERAL EMBOLISM (Vascular disorders) | 2 (2) | 0 (0)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes